CLINICAL TRIAL: NCT01851395
Title: Inpatient Hospice With Procurement of Tissue on Expiration in Thoracic Malignancies, Bladder Cancer, Ovarian Cancer, Epithelial Cancer and Patients Treated With an Adoptive Cellular Therapy
Brief Title: Rapid Autopsy and Procurement of Cancer Tissue
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130131; 13-C-0131
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-30

CONDITIONS: Thymus Tumors; Adoptive Cellular Therapy; Mesothelioma; Genitourinary Cancers; Lung Cancers
Keywords: Palliative; Tumor Heterogeneity; Genomic and Proteomic Alterations; Deep Sequencing and Global Analysis; Clonal Evolution; Natural History
MeSH Terms: conditions — Thymus Neoplasms; Mesothelioma; Urogenital Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1/Thoracic: Patients with histologically or cytologically confirmed metastatic NSCLC, SCLC, EPCC, pNET, thymic epithelial tumor (thymoma, thymic carcinoma) or mesothelioma
- 2/Genitourinary: Patients with genitourinary malignancies
- 3/ACT: Patients treated with an adoptive cellular therapy
- 4/Ovarian: Patients with ovarian cancer
- 5/Epithelial: Patients with breast, colorectal, pancreatic, stomach or biliary cancer.

SUMMARY:
Background:

- Individuals with cancer of the lung, chest cavity, ovary, or bladder, as well as patients who have been treated with adoptive cell therapy unfortunately commonly succumb to their disease. Some agree to donate their bodies to cancer research that may help the medical community better understand these diseases. Studies of cancer tumor tissue obtained soon after death may be used to answer questions about the origins, progression, and treatment of cancer. Researchers want to conduct a study that involves planned collection of cancer tumor tissue shortly after death. To do so, they will arrange to provide inpatient hospice care for people with lung cancer, ovarian cancer, bladder cancer, or patients who have been treated with adoptive cell therapy.

<TAB>

Objectives:

- To collect cancer tissue biopsy samples as soon as possible after death.

Eligibility:

- Individuals who have cancer of the lung, chest cavity, ovary, or bladder, or those who have been treated with adoptive cell therapy and are planning to receive end-of-life hospice care are eligible to participate.

Design:

* Participants will agree to receive inpatient hospice care at the National Institutes of Health Clinical Center. Full details on end-of-life care preference will be acknowledged.
* An autopsy will be performed at the clinical center within 3 hours of death. Tumor tissue will be collected from the primary site of cancer and from any areas of the body to which the cancer has spread.
* Participants will not receive further cancer treatments as part of this study. This is a tissue collection study only.

DETAILED DESCRIPTION:
Background:

* Despite being the leading cause of cancer-related death worldwide, there is only limited knowledge of tumor heterogeneity in lung cancer. There is also limited knowledge of tumor heterogeneity of other less common thoracic malignancies, such as thymic epithelial tumors and mesothelioma. The extent and causes of intra-tumor and inter-metastatic heterogeneity in thoracic malignancies and how they compare to other tumor types is of utmost importance in managing lung cancer. Newer approaches of treating malignancies by targeting immune cells or tumor microenvironment are emerging. Adoptive cellular therapy (ACT) is one such approach. How this therapy affects individual metastatic sites and specific clones of tumor cells is poorly understood.
* Little is known about the clonal architecture of advanced, heavily-treated urothelial carcinoma or the dynamics that lead to metastasis and chemotherapy and immunotherapy resistance. Urothelial carcinomas have a high somatic mutation rate similar to that of non-small cell lung cancer and melanoma. Urothelial carcinoma tumors are extremely heterogenous and the extent of heterogeneity post treatment is an important area of research that should be further explored. Understanding the genetic and clonal evolution of urothelial carcinoma tumors will eventually help guide management of treatment-resistant metastatic tumors.
* Ovarian carcinoma is frequently associated with poor clinical outcome and metastatic disease. Although metastatic processes are becoming more understandable, the genomic landscape and metastatic progression in ovarian cancer has not been elucidated. Despite prior efforts such as The Cancer Genome Atlas (TCGA) and other analyses that were predominantly focused on samples from patients who had upfront debulking surgery, an understanding of the molecular and cellular heterogeneity of ovarian cancer based on highly clinically annotated samples is lacking.
* There is a major need for effective immunotherapies against the common epithelial cancers that account for the vast majority of cancer deaths. Even for lung cancer, where checkpoint inhibition has some efficacy, the majority of these patients do not respond. One option to address these cancers is the adoptive transfer of tumor reactive T-cells (Adoptive Cell Therapy, ACT), which has already demonstrated durable complete cancer regression in a few cases. This approach requires ways to either enrich for tumor-reactive T-cells from tumor infiltrating lymphocytes (TIL) or to rapidly clone mutation-reactive T-cell receptors and use them to engineer T-cell populations for administration. The T-cell response to tumor specific mutations (neoantigens) is highly patient specific and greatly affected by tumor heterogeneity. Developing better ways to d select TIL and TCR for clinical use are needed to advance ACT.
* Tumor heterogeneity can be evaluated in a comprehensive manner by deep sequencing and globally analyzing genomic and proteomic alterations of simultaneous core biopsies from several areas of the primary tumor and metastases. These analyses correlated with clinical outcomes can further the evaluation of tumor heterogeneity. However, such studies are not feasible in a clinical setting.
* Tissue procurement by rapid autopsies provides an effective way for such an investigation.

Objectives:

- Procure primary and metastatic tissue of thoracic malignancies, ovarian cancer, bladder cancer, epithelial cancer (breast, colorectal, pancreatic, stomach or biliary cancers) and from patients treated with an ACT shortly after death, to investigate tumor heterogeneity and immune microenvironment intratumorally, between paired primary and metastatic sites, and among inter-metastatic tumors using integrated genomic, immunologic and proteomic analysis.

Eligibility:

- Adult patients with metastatic non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), extrapulmonary small cell cancer (ESCC), pulmonary neuroendocrine tumor (pNET), thymic epithelial tumor, mesothelioma, bladder cancer (including urothelial carcinoma and other rare bladder or kidney histology), ovarian cancer, epithelial cancer and patients treated with an ACT, with no expected chance of cure and an expected survival of less than 3 months.

Design:

* The accrual ceiling for the study will be set at 275 in order to account for subjects that for whatever reason do not undergo autopsy.
* Patients will be admitted for inpatient hospice when an investigator evaluates that death is clinically imminent.
* Upon expiration, rapid autopsy will be performed and tissue will be obtained from the primary tumor site, if identifiable, and multiple metastatic sites to assess tumor heterogeneity and immune microenvironment using deep sequencing and global genomic and proteomic analyses.
* Archival tissue from patients, if available, will be used to evaluate these changes from several stages of tumor progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed metastatic NSCLC, SCLC, EPCC, pNET, thymic epithelial tumor (thymoma, thymic carcinoma) or mesothelioma confirmed by the NCI Laboratory of Pathology. Patients with bladder cancer (including urothelial carcinoma and other rare bladder or kidney histology), ovarian cancer, epithelial cancers (breast, colorectal, pancreatic, stomach and biliary cancers) and malignancies previously treated with an ACT are also eligible.
* Age >= 18 years.
* Incurable disease or terminal diagnosis.
* Patients or legally authorized representative (LAR) must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must provide valid written designation of an assigned Durable Power of Attorney (DPA). If one is not available, an LAR must be assigned.
* Patients and their legal next of kin must agree to a Do Not Resuscitate (DNR) order and agree to Consent for Autopsy as part of the end-of-life care plan.

EXCLUSION CRITERIA:

* Women known to be pregnant (known positive pregnancy test, although such testing is not required for enrollment) are excluded.
* Known HIV-positive patients will be excluded (although HIV testing is not required for enrollment) because of the potential for contamination of tissue.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected primarily from the CC medical oncology clinic setting.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2013-12-30 (Actual); Primary Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Tumor heterogeneity | Death
  Both intratumor and between paired primary and metastatic site, using integrated genomic and proteomic analysis.

SECONDARY OUTCOMES:
Genetic alterations | completion of study
  To compare genetic alterations of autopsied tissue with archival tissue from primary and metastatic sites when available, to evaluate heterogeneity between primary and metastatic sites and at two different times during tumor evolution.-Compare genomic alterations in tumor tissue with those identified in isolated circulating tumor cells from blood obtained during the short hospital stay before death.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0131.html